CLINICAL TRIAL: NCT04222296
Title: Clinical Evaluation of Outcomes With Hearing Aid Parameters Designed for Adults With Severe-profound Hearing Loss and Unilateral Cochlear Implants in Bimodal (Cochlear Implant and Contralateral Hearing Instrument), CROS (Contralateral Routing of Signals) and Bilateral Amplification Strategies
Brief Title: Bimodal, CROS and Severe Profound Hearing Loss Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Advanced Bionics AG (Industry)
Responsible Party: Principal Investigator, James Tysome, Consultant ENT and Skull Base Surgeon, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/EE/0160
Record Dates: First submitted 2019-01-23; First posted 2020-01-09 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Cochlear Implant; Severe-Profound Hearing Loss; Hearing Loss, Bilateral; Hearing Loss, Cochlear
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cochlear Implant and Hearing Aid (Other): Comparing performance of conventional hearing aid fitting to Phonak's Bimodal Fitting formula using the Phonak Naida Link hearing aid. All patients are tested in a bimodal (hearing aid plus cochlear implant) setup. Initial tests are completed with the Advanced Bionics Naida Q70 or Q90 sound processor and the patient's own hearing aid. In this arm, a patient's own hearing aid is replaced with the Phonak Naida Link hearing aid to test if there is a benefit.
  Interventions: Device: Fitting strategy of cohlear implant of hearing aid
- Cochlear Implant alone (Other): To determine if the addition of a contralateral routing of signal (CROS) microphone on the un-implanted ear improves performance. Baseline tests are completed with Advanced Bionics Naida Q70 or Q90 sound processors. Patients are then given the Phonak Naida Link CROS aid to test if there is a benefit.
  Interventions: Device: Fitting strategy of cohlear implant of hearing aid
- Hearing Aid and Hearing Aid (Other): Comparing performance of conventional hearing aid fitting to a modified signal processing strategy more aligned with how a cochlear implant manages sound. All patients are tested initially with their own hearing aids to obtain a baseline measurement. Patients are then fitted with a modified Phonak hearing aid to determine if performance improves.
  Interventions: Device: Fitting strategy of cohlear implant of hearing aid

INTERVENTIONS:
Device: Fitting strategy of cohlear implant of hearing aid — To determine whether new hardware and fitting strategy provides better sound quality or ease of use than generic hardware and fitting methods

SUMMARY:
The study will involve the comparison of three groups with severe-profound hearing loss. Patients with a Cochlear Implant only, patients with a cochlear implant and Hearing Aid, and finally patients with two hearing aids.

This will enable a comparison of standard fitting protocols against the new rationale using the same devices. Devices used for patients in all 3 groups are now available in standard of care, and can be kept afterwards should the patients wish.

DETAILED DESCRIPTION:
The study will involve three groups of 20 patients per group. This first is experienced adult bimodal users of the AB system who have usable contralateral residual hearing. A clinical baseline and three research conditions will be evaluated.

The Naida CI Link HA (Link) will be fitted, tested and then optimised using a special bimodal fitting formula. Subjects will be allowed three months to acclimatize and will then be retested. The second research condition will evaluate the fully integrated bimodal system, where the microphone signals from CI and HA are shared and a bilateral beamformer is formed. A third intervention will involve modifying the CI settings to minimize the mis-match between frequencies delivered via the CI.

A second group with no aidable hearing on their non-implanted ear will also be studied. A contralateral routing of signal (CROS) device will send sounds on the non-implanted side. Tests will be made with and without CROS, as well as with directional microphone settings.

Finally as a control group, bilateral HA users will be tested with the similar HA fitting as used for the bimodal group.

This will enable a comparison of standard fitting protocols against the new rationale using the same devices.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Consistent unilateral user of an Advanced Bionics cochlear implant and a contralateral hearing aid for at least 6 months, ideally 12 months, and Bilateral severe to profound hearing loss (meeting NICE criteria for implantation-2009). (group 1)
* Consistent unilateral user of an Advanced Bionics cochlear implant for at least 6 months and ideally 12 months, with no useful contralateral hearing (group 2)
* Consistent user of bilateral hearing aids for at least six months (group 3) and bilateral severe profound hearing loss (80dB or worse at 2000 and 4000 Hz with speech discrimination of at least 50% IHR sentences live voice at 60dBA)
* First language English
* Post-lingual onset of severe to profound hearing loss
* No other handicaps that would interfere with participation in the study in the opinion of the Principle Investigator

Exclusion Criteria:

* Unstable cochlear implant or hearing aid fitting
* Using medication in an intermittent manner that might influence hearing levels
* Cognitive or psychological challenges that might lead to variations in attention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Sound Processing parameters | 24 months
  ASSE score

CONTACTS AND LOCATIONS:
Overall Officials: James R Tysome, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided